CLINICAL TRIAL: NCT07361289
Title: A Single-Arm Observational Study to Assess the Real-World Effectiveness of Mavacamten in Adult Patients With Obstructive Hypertrophic Cardiomyopathy in China
Brief Title: A Study to Assess the Real-World Effectiveness of Mavacamten in Adult Patients With Obstructive Hypertrophic Cardiomyopathy in China
Acronym: SOAR-HCM
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1210
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Obstructive hypertrophic cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cohort 1: Participants with symptomatic obstructive hypertrophic cardiomyopathy (oHCM) receiving mavacamten
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — According to the product label

SUMMARY:
The purpose of this study is to assess the effectiveness of mavacamten treatment in Chinese adults with symptomatic obstructive hypertrophic cardiomyopathy (HCM) in real-world clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years (participants enrolled retrospectively: at the time of initial mavacamten prescription), irrespective of gender.
* Diagnosed with obstructive hypertrophic cardiomyopathy (HCM) consistent with current American College of Cardiology Foundation/American Heart Association, European Society of Cardiology, and Chinese guidelines for diagnosis and treatment of patients with hypertrophic cardiomyopathy, i.e., satisfy criteria below:

  * Has unexplained left ventricular (LV) hypertrophy with non-dilated ventricular chambers in the absence of other cardiac (e.g., hypertension, aortic stenosis) or systemic disease and with maximal LV wall thickness ≥ 15 mm (or ≥ 13 mm with positive family history of hypertrophic cardiomyopathy) in the most recent medical record within 3 months prior to enrollment, and
  * Peak left ventricular outflow tract (LVOT) gradient ≥ 30 mmHg at rest or with provocation in the most recent medical record within 3 months prior to enrollment as assessed by echocardiography.
* Has documented left ventricular ejection fraction (LVEF) ≥ 55%, as measured by resting transthoracic echocardiography (TTE) in the most recent medical record within 3 months prior to enrollment.
* New York Heart Association (NYHA) class II or III symptoms in the most recent medical record within 3 months prior to enrollment.
* Participants who have initiated mavacamten (for whom enrolled retrospectively) or are scheduled to initiate mavacamten (for whom enrolled prospectively) based on clinical therapeutic needs.
* For participants enrolled retrospectively, must have traceable essential baseline information (including age, gender, resting LVOT peak gradient, Valsalva LVOT peak gradient, LVEF, indices of cardiac structure, systolic and diastolic function, cardiac biomarkers, NYHA functional class) and critical data (including resting and Valsalva LVOT gradient, LVEF, cardiac structure, systolic and diastolic function, dose of mavacamten) at key follow-up time points that have been completed.
* Voluntary sign informed consent form.

Exclusion Criteria:

* Known HCM phenocopy disease (e.g., Fabry disease, amyloidosis).
* Participants who are expected to undergo major cardiac surgery during the study.
* Prior treatment of obstructive HCM with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA] or septal radiofrequency ablation) within 6 months prior to enrollment (participants enrolled retrospectively: within 6 months prior to initial mavacamten prescription); participants with an unsuccessful myectomy or percutaneous ASA or septal radiofrequency ablation performed >6 months prior to enrollment (participants enrolled retrospectively: within 6 months prior to initial mavacamten prescription) may be enrolled.
* Currently treated with disopyramide or ranolazine (within 14 days prior to enrollment [participants enrolled retrospectively: within 14 days prior to initial mavacamten prescription]) or participants who are expected to be taking disopyramide, ranolazine, verapamil in combination with β-receptor blockers, or diltiazem in combination with β-receptor blockers during the study.
* Presence of other diseases that may affect completion of 96 weeks follow-up as assessed by the investigator.
* Participants who are using or are expected to be using moderate to strong CYP2C19 inhibitors/inducers, or strong CYP3A4 inhibitors, moderate to strong CYP3A4 inducers during the study.
* Participants who are participating in other interventional clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults diagnosed with symptomatic obstructive hypertrophic cardiomyopathy that have received mavacamten treatment in China
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2028-08-22 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Valsalva left ventricular outflow tract (LVOT) gradient | Week 48, Week 96
Change from baseline in resting valsalva left ventricular outflow tract (LVOT) gradient | Week 48, Week 96

SECONDARY OUTCOMES:
Change from baseline in New York Heart Association (NYHA) class | Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, and Week 96
Number and proportion of participants with a resting/provoked left ventricular outflow tract (LVOT) gradient < 30/50 mmHg | Week 12, Week 36, Week 48, Week 72, and Week 96
Number and proportion of participants achieving complete response (defined as all left ventricular outflow tract (LVOT) gradients < 30 mmHg and New York Heart Association (NYHA) Class I) | Week 12, Week 36, Week 48, Week 72, and Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- China (15):
  - Local Institution - 0008, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Local Institution - 0002, Beijing, Beijing Municipality
  - Local Institution - 0009, Guangzhou, Guangdong
  - The Second Afilliated Hospital of Hebei Medical University, Jiazhuang, Hebei
  - Local Institution - 0003, Harbin, Heilongjiang
  - Local Institution - 0007, Zhengzhou, Henan
  - Local Institution - 0015, Suzhou, Jiangsu
  - Local Institution - 0004, Changchun, Jilin
  - Local Institution - 0005, Dalian, Liaoning
  - Local Institution - 0013, Xi'an, Shan3xi
  - Local Institution - 0012, Chengdu, Sichuan
  - Local Institution - 0006, Hangzhou, Zhejiang
  - Local Institution - 0010, Jinan
  - Local Institution - 0011, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts